CLINICAL TRIAL: NCT03982862
Title: Intralesional Injection of Steroids and/or Botulinum Toxin Type A in Hypertrophic Scars and Keloids for Pain Improvement
Brief Title: Botulinum Toxins Intralesional Injection for Scar Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Sheng-Hua Wu, Attending Physician, anesthesiology, Kaohsiung Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20180062
Record Dates: First submitted 2019-06-09; First posted 2019-06-12 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Scar Keloid; Hypertrophic Scar
Keywords: Botulinum toxin type A; Triamcinolone; scar pain; scar itch
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic | interventions — Triamcinolone; Steroids; Lidocaine; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): 0.9% Normal saline 0.1 ml +Triamcinolone 4mg diluted to 0.1 ml + 0.1ml 2% Xylocaine per 1cm2 scar volume
  Interventions: Drug: Triamcinolone; Drug: Lidocaine
- botox group (Experimental): 4U Botox® diluted to 0.1 ml + Triamcinolone 4mg diluted to 0.1 ml + 0.1ml 2% Xylocaine per 1 cm2 scar volume
  Interventions: Drug: Triamcinolone; Drug: Lidocaine; Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Triamcinolone — Triamcinolone 4mg diluted to 0.1 ml
  Other Names: steroid
Drug: Lidocaine — 0.1ml 2% Xylocaine
  Other Names: Xylocaine
Drug: Botulinum toxin A — 4U Botox® diluted to 0.1 ml
  Other Names: botox
  Arms: botox group

SUMMARY:
Botulinum toxins has been approved by the FDA to treat chronic migraine. Botox had been shown to inhibiting the release of inflammatory mediators and peripheral neurotransmitters from sensory nerve to treat neuropathic pain. In the clinical practice, botox indeed effect in scar pain. However, investigators need well controlled study to prove this finding and assess the improvement of scar appearance.

DETAILED DESCRIPTION:
After surgery or trauma, scar tissues would form during the healing process. However, hypertrophic scars and keloids might happen to some patients, both of which are often pruritic and erythematous. Besides, the markedly elevated tumor-like appearance usually brings much concern to patients. Moreover, significant pain or discomfort could happen to keloids. Various treatment strategies were mentioned but without a solid solution to all of the scars. Investigators hope to evaluate the differences of scar volume, appearance and symptoms (itching and pain) in participants receiving simultaneous intralesional injection of Botulinum toxin type A and/or steroids. Besides, side effects would also be recorded. Investigators hope to establish a more effective intralesional injection therapy for participatns suffering from hypertrophic scars and keloids.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have visible hypertrophic scars or keloids over three months after trauma or surgery.
2. Patients have symptoms of pain, itching or erythema.

Exclusion Criteria:

1. Patients had either Botulinum toxin type A or Triamcinolone intralesional before in the same scar
2. The scar size is larger than 10 cm2
3. Immunocompromised status
4. Systemic infection status
5. Allergic to Botulinum toxin type A or steroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Scar pain relief | Change from baseline scar pain during 16 weeks after drug injection
  assessed by score 0,1,2 (0: no pain, 1: sometimes feel pain, 2: need medication)
scar appearance | Change from baseline scar appearance during 16 weeks after drug injection
  assessed by vancouver scar scale(vascularity, pigmentation, pliability, height)
itch | Change from baseline itch sensation during 16 weeks after drug injection
  assessed by score 0,1,2 (0: no itch, 1: sometimes feel itch, 2: need medication)

CONTACTS AND LOCATIONS:
Overall Officials: Shu Hung Huang, MD, PHD, Study Director — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan